CLINICAL TRIAL: NCT03031704
Title: French Register of Duodenal Adenomas Characterization and Evaluation of Endoscopic Mucosectomy
Acronym: MUCO-DUO
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Other Study IDs: 2016-27
Record Dates: First submitted 2017-01-23; First posted 2017-01-26 (Estimated); Last update posted 2017-01-26 (Estimated); Status verified 2017-01

CONDITIONS: Duodenal Adenoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Endoscopic mucosectomy
  Interventions: Procedure: Endoscopic mucosectomy

INTERVENTIONS:
Procedure: Endoscopic mucosectomy — Performing adenoma resection through standardized endoscopic mucosectomy of duodenal adenoma.

SUMMARY:
Sporadic duodenal adenomas are rare. As they are highly pre neoplastic, they should be removed and endoscopic mucosectomy is recommended during digestive endoscopy. However, this technique, albeit less dangerous than surgery, is associated with complications such as haemorrhages, perforations, and more relapse than that can be observed for colorectal adenomas. As no prospective data have been published this French multicenter study aim to analyze results of this technique under standardized and secured procedure.

All investigators are expert in therapeutic endoscopy in tertiary centers and are member of a group of clinical researcher involved in that field (" GRAPHE " (Groupe de Recherche et d'Action des Praticiens Hospitaliers en Endoscopie interventionnelle). Results are highly expected among the international society of gastroenterologists who need to confirm the efficacy of endoscopy and define optimal conditions for performing adenomas resection in this location Primary End Point is the two years recurrence rate. Secondary End Points are frequency and type of complication after standardized endoscopic mucosectomy of duodenal adenomas, frequency and type of complications after a second endoscopic mucosectomy and patient's characteristics Patients with sporadic duodenal adenomas larger than 5 mm requiring endoscopic mucosectomy will be included. Non-inclusion criteria concern patients with previous endoscopic resection, lesion involving the major papilla, sub mucosal lesions, familial adenomatous polyposis and use of antiplatelet agent during the five last days.

Hundred and twenty patients will be included and followed 2 years after mucosectomy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with sporadic duodenal adenomas larger than 5 mm requiring endoscopic mucosectomy

Exclusion Criteria:

* patients with previous endoscopic resection,
* patients prsenting lesion involving the major papilla, sub mucosal lesions
* patient with familial adenomatous polyposis
* patient undergoing use of antiplatelet agent during the five last days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with sporadic duodenal adenomas larger than 5 mm requiring endoscopic mucosectomy will be included
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2017-01-09 (Actual); Primary Completion 2021-01-09 (Estimated); Study Completion 2022-01-09 (Estimated)

PRIMARY OUTCOMES:
Number of recurrence after surgery | 2 yeras

CONTACTS AND LOCATIONS:
Overall Officials: Urielle DESALBRES, Study Director — Assistance Publique Hôpitaux de Marseille
Locations (1):
- Assistance Publique Hôpitaux de Marseille, Marseille, France

IPD SHARING:
Plan to Share IPD: No